CLINICAL TRIAL: NCT06872645
Title: Exploring Water-free Sodium Storage
Acronym: NOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000039499; 1R01DK138155 (NIH)
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Peritoneal Dialysis, Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Glucose; Water

STUDY DESIGN:
Intervention Model Description: Randomized, blinded crossover study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 5% dextrose peritoneal dialysis, 2-hour dwell (Experimental): Individuals will receive up to 2 liters of 5% dextrose for peritoneal dialysis during up to a 2-hour dwell for 5 days
  Interventions: Drug: 5% Dextrose/Water
- 1.5% dextrose peritoneal dialysis, 2-hour dwell (Active Comparator): Individuals will receive up to 2 liters of 1.5% dextrose for peritoneal dialysis during up to a 2-hour dwell for 5 days
  Interventions: Drug: 1.5% standard PD fluid

INTERVENTIONS:
Drug: 5% Dextrose/Water — Patients will be randomized to undergo up to two-hour dwell with 5% dextrose in sterile water for 5 days
  Arms: 5% dextrose peritoneal dialysis, 2-hour dwell
Drug: 1.5% standard PD fluid — Patients will be randomized to undergo up to two-hour dwell with 1.5% standard PD fluid for 5 days
  Arms: 1.5% dextrose peritoneal dialysis, 2-hour dwell

SUMMARY:
The overarching goal of this proposal is to definitively establish if acute water free Na storage and release occurs, if the amount stored/released is of a quantity that is physiologically relevant, and if the location is intracellular vs. extracellular.

DETAILED DESCRIPTION:
This study is designed as a an ultra-rigorous inpatient balance study. The main purpose of the study is to determine if significant mobilizable non- extracellular volume (ECV) Na storage occurs in humans. This is a randomized, blinded crossover study. Patients will be randomized to Na free 5% dextrose solution or 1.5% standard peritoneal dialysis (PD) fluid (Dianeal 1.5% low calcium PD solution with standard 132 mmol/L Na and osmolarity of 344 mOsmol/L) and will receive treatment for 5 days, following a 6 week wash out patient will return to undergo 5 days of alternate therapy.

ELIGIBILITY:
Inclusion Criteria:

* ESRD Patients actively undergoing PD with a reliably functioning PD catheter
* Systolic blood pressure > 130 mmHg
* Serum sodium >135 mmol/L
* daily urine output < 400ml
* stable PD prescription for at least 2 months without requirement of 4.25% glucose PD solution
* PD vintage of at least 6 months
* Euvolemic as defined by the patient at their dry weight and free of any signs or symptoms of volume overload, per referring nephrologist

Exclusion Criteria:

* Poorly controlled diabetes with hemoglobin A1C>9%
* 1 or more episodes of peritonitis in the previous 6 months or active infection of the peritoneal dialysis catheter
* Anemia with hemoglobin <8g/dL
* Inability to give written informed consent or follow study protocol.
* Urinary incontinence
* Body weight < 60kg
* gastrointestinal disease that causes diarrhea or expectation of sodium losses in stool.
* use of amiodarone in the last 6 months (which will interfere with tissue iodine ascertainment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Water free Na removal over the 5-day intervention | Daily for 5 days
  Water free Na removal will be calculated as [Water Free Na= ((ΔTBW (L) * serum Na (mmol/L)) - Na balance (mmol)]. This will be compared between 5% dextrose Na removal period and 1.5% dextrose standard PD neutral Na balance period

OTHER OUTCOMES:
Change in total extracellular Na and osms | Day 1 and day 5
  Change in total extracellular Na and osms will be calculated as [Change ECV Na = {ECV (L) * serum Na (mmol/L at baseline} - {ECV (L) * serum Na (mmol/L) after dwell).
  The same approach will be done for osms

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No